CLINICAL TRIAL: NCT00543686
Title: A Randomised Controlled Open-Label Phase IV Mono Centre Study to Compare the Response Profiles of Montelukast Versus Fluticasone in Children With Pre-School Asthma
Brief Title: Leukotriene Receptor Antagonists or Steroids in Pre-School Asthma
Acronym: LOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof Stefan Zielen, Goethe University, Childrens Hospital, Dpt of Pulmonology, Frankfurt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 165/07/FFM
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
Keywords: Pre-School Asthma; Responder Profiles; Fluticasone; Montelukast; Leukotriene; Children with Pre-School Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Montelukast
  Interventions: Drug: Montelukast
- 2 (Active Comparator): Fluticasone
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Montelukast — Intake of Montelukast
  Arms: 1
Drug: Fluticasone — Intake of Fluticasone
  Arms: 2

SUMMARY:
Explorative comparison of montelukast with inhaled steroids (fluticasone) to estimate responder profiles, in terms of symptom scores, rescue medication, increase of FEV1, in correlation to presence of allergy, bronchial hyperreactivity (PD20), exhaled NO, excretion of leukotrienes, response to RABA and laboratory parameters in patients with pre-school asthma i.e. asthma phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 4 -6 years
* Diagnosis of mild intermittent bronchial asthma (Step I-II) in the past 6 - 12 months as stated by the investigator:
* Use of inhaled beta-2-agonists < 1/week (max 3 puff /d)
* Exacerbation-free interval > 4 weeks prior to visit 1
* The written informed consent of parents after received written and oral information about the aim, purpose and risks of the study must be present

Exclusion Criteria:

* Asthma severity ≥ Step 2
* Severe concomitant diseases
* Suspected non-compliance
* age below 4 and age above 7 years
* last study participation < 30 days

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the number of responders with a very good asthma symptom control defined as requiring no rapid acting beta agonist (RABA) between the 2. and 6th week of intervention (end of trial)

SECONDARY OUTCOMES:
the number of patients requiring at least five times RABA between the 2. and 6th week, the number of patients with an increase of FEV1 7.5%, the symptom score, symptom free days, rescue medication, presence of allergy RAST > 2, concentration of eNO, PD20

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof. Dr., Principal Investigator — Johann Wolfgang Goethe-University Frankfurt, Zentrum für Kinderheilkunde I, Haus 32, Abt. Pneumologie
Locations (1):
- Goethe University, Department of Pulmonology, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Zielen S, Christmann M, Kloska M, Dogan-Yildiz G, Lieb A, Rosewich M, Schubert R, Rose MA, Schulze J. Predicting short term response to anti-inflammatory therapy in young children with asthma. Curr Med Res Opin. 2010 Feb;26(2):483-92. doi: 10.1185/03007990903485148. PMID 20001651